CLINICAL TRIAL: NCT06522217
Title: Prosthetic Rehabilitation of Lip and Palate Deformaties in Neonates Using Two Different Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdallah, lecturer of removable and maxillofacial prosthodontics, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP-12-18
Record Dates: First submitted 2024-07-11; First posted 2024-07-26 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-07

CONDITIONS: Evaluation
Keywords: nasoalveolar molding; digital nasoalveolar molding; complete unilateral cleft lip and palate

STUDY DESIGN:
Intervention Model Description: 2 groups : Group A receiving conventional nasoalveolar molding appliance and Group B receiving CAD NAM
Who Masked: Participant, Care Provider
Masking Description: starting 2 conventional then 2 CAD NAM patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Group A (Active Comparator): 10 neonates receiving conventional nasoalveolar molding appliances
  Interventions: Device: nasoalveolar molding appliance
- Digital Group B (Active Comparator): 10 neonates receiving CAD- nasoalveolar molding appliances
  Interventions: Device: digital nasoalveolar molding appliance

INTERVENTIONS:
Device: nasoalveolar molding appliance — making impression then make the conventional lab procedures for group A for the production of conventional appliances
  Arms: Conventional Group A
Device: digital nasoalveolar molding appliance — group B scanning the model and designing the appliances on 3shap and 3d printing the appliances
  Arms: Digital Group B

SUMMARY:
This study was conducted to compare the use of conventional nasoalveolar molding appliances and the use of digitally designed and produced nasoalveolar molding appliances in rehabilitating neonates born with unilateral complete cleft lip and palate.

DETAILED DESCRIPTION:
For this prospective study, twenty newborns with non-syndromic complete unilateral cleft lip and palate were referred from the Outpatient Clinics of several pediatric surgeons and obstetricians to the Department of Prosthodontics -Faculty of Dentistry - Tanta University.

Inclusion criteria:

* Age range from 2-3 weeks after birth.
* Only the Non-syndromic unilateral cleft lip and palate neonates.
* Newborn infants without any surgical intervention.

Exclusion criteria:

* Patients with the life threatening syndromes.
* Respiratory difficulties are not considered for presurgical treatment.
* Uncooperative guardians.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 2-3 weeks after birth.
* Only the Non-syndromic unilateral cleft lip and palate neonates.
* Newborn infants without any surgical intervention.

Exclusion Criteria:

* Patients with the life threatening syndromes.
* Respiratory difficulties are not considered for presurgical treatment.
* Uncooperative guardians.

Ages: 2 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
intraoral measurements | 3 -4 months
  measuring 2 points the first is the intersegmental distance in (mm) and the second is the alveolar width in (mm)
extraoral measurements | 3-4 months
  * Nostril height in (mm)
  * Nasal dome height in (mm)
  * Columella height in( mm)
  * Nostril basal width in (mm)
  * Nostril width in (mm)

CONTACTS AND LOCATIONS:
Overall Officials: hoda amin rashad, phd, Principal Investigator — tanta university faculty of dentistry
Locations (1):
- Faculty of Dentistry -Tanta university, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No